CLINICAL TRIAL: NCT03349788
Title: Randomized Controlled Trial: Clinical Value of Preserving Left Colic Artery in Laparoscopic Radical Rectectomy
Brief Title: Clinical Value of Left Colic Artery in Laparoscopic Radical Rectectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ShanghaiMISC-LCA
Record Dates: First submitted 2017-11-09; First posted 2017-11-22 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-11

CONDITIONS: Overall Survival; Postoperative Complications
Keywords: Left colic artery; Laparoscopic Surgery; Anterior resection of rectum; Rectum cancer
MeSH Terms: conditions — Postoperative Complications; Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LCA-nP (Experimental): The group underwent laparoscopic radical rectectomy without preserving left colic artery. In IMA group, the dissecting based on TME is performed without preserving left colic artery. Surgeon should dissect the lymph nodes and ligated the vessel in the root of inferior mesenteric artery.
  Interventions: Procedure: LCA-nP
- LCA-P (Active Comparator): The group underwent laparoscopic radical rectectomy with preserving left colic artery. In LCA group, the dissecting based on TME is performed with preserving left colic artery. The relationship of inferior mesenteric artery, inferior mesenteric vein and LCA should be identified and ligated separately without LCA.
  Interventions: Procedure: LCA-P

INTERVENTIONS:
Procedure: LCA-nP — The group underwent lapaoroscopic radical rectectomy without preserving left colic artery.
  Arms: LCA-nP
Procedure: LCA-P — The group underwent lapaoroscopic radical rectectomy with preserving left colic artery.
  Arms: LCA-P

SUMMARY:
Colorectal cancer is one of the most common tumors in Asia. According to the recent research, surgical procedure could provide more treatment benefit in rectal cancer. Therefore, it was consider that important to standardized and improved the surgical procedure for rectal cancer. With the development of anatomical technique, minimally surgery with laparoscopy had become the trend for surgical treatment. There were several studies has been done to evaluate the safety and feasibility of laparoscopic surgery. In order to achieve better surgical outcome and reduce operative complications, the investigators design stratified randomization, double blinded, muti - center clinical trail to investigate the value of left colic artery in laparoscopic radical rectectomy.

ELIGIBILITY:
Inclusion Criteria:

* Aged more then 18 years old;
* Diagnosed as rectal cancer with colonoscopic biopsy;
* Without metastasis;
* No Invasion of surrounding tissues;
* Limited operation;
* Underwent laparoscopic radical proctectomy(L-Dixon);
* BMI 18~30kg/m2;
* Without multiple primary tumors;
* Sign on the Medical informed Consent.

Exclusion Criteria:

* Simultaneous or simultaneous multiple primary colorectal cancer;
* Preoperative imaging examination results show: (1) Tumor involves the surrounding organs and combined organ resection need to be done; (2)distant metastasis; (3)unable to perform R0 resection;
* History of any other malignant tumor in recent 5 years;
* Patients need emergency operation;
* Not suitable for laparoscopic surgery;
* Women during Pregnancy or breast feeding period;
* Informed consent refusal

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 3 years

SECONDARY OUTCOMES:
The rate of postoperative coml[ications and mortality | 30 days
3 years overall survival | 3 years
The rate of local and distant recurrence | 3 years
The rate of LN.253 metastasis | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Minhua Zheng, PhD, Study Director — Ruijin Hospital
Locations (1):
- Shanghai Ruijin Hospttal, Shanghai, Sahgnhai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lange MM, Buunen M, van de Velde CJ, Lange JF. Level of arterial ligation in rectal cancer surgery: low tie preferred over high tie. A review. Dis Colon Rectum. 2008 Jul;51(7):1139-45. doi: 10.1007/s10350-008-9328-y. Epub 2008 May 16. PMID 18483828
- [Result] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Result] Brenner H, Kloor M, Pox CP. Colorectal cancer. Lancet. 2014 Apr 26;383(9927):1490-1502. doi: 10.1016/S0140-6736(13)61649-9. Epub 2013 Nov 11. PMID 24225001
- [Result] Deijen CL, Velthuis S, Tsai A, Mavroveli S, de Lange-de Klerk ES, Sietses C, Tuynman JB, Lacy AM, Hanna GB, Bonjer HJ. COLOR III: a multicentre randomised clinical trial comparing transanal TME versus laparoscopic TME for mid and low rectal cancer. Surg Endosc. 2016 Aug;30(8):3210-5. doi: 10.1007/s00464-015-4615-x. Epub 2015 Nov 4. PMID 26537907
- [Result] Uehara K, Yamamoto S, Fujita S, Akasu T, Moriya Y. Impact of upward lymph node dissection on survival rates in advanced lower rectal carcinoma. Dig Surg. 2007;24(5):375-81. doi: 10.1159/000107779. Epub 2007 Aug 4. PMID 17785983
- [Result] Cirocchi R, Trastulli S, Farinella E, Desiderio J, Vettoretto N, Parisi A, Boselli C, Noya G. High tie versus low tie of the inferior mesenteric artery in colorectal cancer: a RCT is needed. Surg Oncol. 2012 Sep;21(3):e111-23. doi: 10.1016/j.suronc.2012.04.004. Epub 2012 Jul 6. PMID 22770982
- [Result] Kim HJ, Kim CH, Lim SW, Huh JW, Kim YJ, Kim HR. An extended medial to lateral approach to mobilize the splenic flexure during laparoscopic low anterior resection. Colorectal Dis. 2013 Feb;15(2):e93-8. doi: 10.1111/codi.12056. PMID 23061515
- [Result] Mari G, Maggioni D, Costanzi A, Miranda A, Rigamonti L, Crippa J, Magistro C, Di Lernia S, Forgione A, Carnevali P, Nichelatti M, Carzaniga P, Valenti F, Rovagnati M, Berselli M, Cocozza E, Livraghi L, Origi M, Scandroglio I, Roscio F, De Luca A, Ferrari G, Pugliese R. "High or low Inferior Mesenteric Artery ligation in Laparoscopic low Anterior Resection: study protocol for a randomized controlled trial" (HIGHLOW trial). Trials. 2015 Jan 27;16:21. doi: 10.1186/s13063-014-0537-5. PMID 25623323
- [Result] Titu LV, Tweedle E, Rooney PS. High tie of the inferior mesenteric artery in curative surgery for left colonic and rectal cancers: a systematic review. Dig Surg. 2008;25(2):148-57. doi: 10.1159/000128172. Epub 2008 Apr 29. PMID 18446037